CLINICAL TRIAL: NCT03466801
Title: The Efficacy of Prednisone Alone and Combination Therapy With Methylprednisolone and Cyclophosphamide in the Treatment of Membranous Nephropathy in Stage I.
Brief Title: The Efficacy of Prednisone and Combination Therapy With Methylprednisolone and Cyclophosphamide on IMN in Stage I.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the clinical significance is little
Sponsor: Wenhu Liu (Other)
Responsible Party: Sponsor-Investigator, Wenhu Liu, Professor, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-P2-172-02
Record Dates: First submitted 2018-01-13; First posted 2018-03-15 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: prednisone alone; methylprednisolone and cyclophosphamide; membranous nephropathy in stage I
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Prednisone; Glucocorticoids; Immunosuppressive Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group prednisone (Experimental): Prednisone was taken 1mg/kg/d(maximum 60mg/d)for 8 weeks to start.Then decreased 5mg every 2 weeks; When reduced to 40mg,reduced 5mg every 4 weeks. When reduced to 20mg, reduced 2.5mg every 8 weeks until the end.
  Interventions: Drug: Prednisone
- Group MP and CTX (Active Comparator): The first month,Methylprednisolone(MP) was injected for 3 days(weight >60kg,500mg/d;<60 kg,300mg/d),and 0.4mg/kg/d for 27 day.The second month,Cyclophosphamide(CTX) orally was 100mg/d for 1 month.And this regimen is repeated for six months.
  Interventions: Drug: MP and CTX

INTERVENTIONS:
Drug: Prednisone — Prednisone was taken for oral administration with dosage of 1mg/kg/d (maximum 60mg/d) by 8 weeks to start.Then reduced Gradually until the end of the experiment.
  Other Names: Glucocorticoid
  Arms: Group prednisone
Drug: MP and CTX — Methylprednisolone(MP) was injected for 3 day(if weight >60kg ,500mg/d<60kg,300mg/d ), methylprednisolone was 0.4mg/kg/d for 27 day.Cyclophosphamide(CTX) orally was 100mg/ d for 1 month.And repeated for six months.
  Other Names: Glucocorticoid and immunosuppressive agents
  Arms: Group MP and CTX

SUMMARY:
Multi-center, prospective, randomized, controlled study to verify the efficacy of prednisone alone and combination therapy with methylprednisolone and cyclophosphamide in the treatment of stage I membranous nephropathy.

DETAILED DESCRIPTION:
Idiopathic membranous nephropathy (IMN) is one of the most common cause of adult nephrotic syndrome. Prednisolone and methylprednisolone are essential drugs for IMN. However, there are no recommendations for the treatment of IMN in China. KDIGO guidelines recommend combination therapy with methylprednisolone and cyclophosphamide as first-line therapy of IMN, but there is a large side effect of cyclophosphamide.There were retrospective study showed that the use of glucocorticoid hormones (including prednisone and methylprednisolone) alone may be effective in patients with membranous nephropathy in Asia, but there is no high quality evidence of evidence-based medicine.The study is a randomized prospective controlled multi-centered trial,to compare the efficacy of prednisone alone and combination therapy with methylprednisolone and cyclophosphamide in the treatment of membranous nephropathy in stage I.

ELIGIBILITY:
Inclusion Criteria:

1. The pathological examination of renal biopsy was consistent with the early idiopathic membranous nephropathy
2. Meeting one of the following three condition：

   * Urine protein quantitation >4g/d,or 50% higher than baseline,RASS blocker treat for 6 months without trend of decrease ②Serious or disabling complications related to nephrotic syndrome ③In the 6-12 months after diagnosis of idiopathic membranous nephropathy, serum creatinine increased by more than 30%, while eGFR eGFR≥25ml/min/1.73m2.And excludeing other causes of renal dysfunction

Exclusion Criteria:

1. Secondary membranous nephropathy
2. Serious complications
3. Considering the effect of cyclophosphamide on the of function of sex gland，all patients with childbearing age or fertility requirement cannot participate in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
nephrotic syndrome remission ( including complete remission and partial remission) | 12 months
  nephrotic syndrome remission ( including complete remission and partial remission)

SECONDARY OUTCOMES:
blood albumin≥30g/L | 12 months
  blood albumin≥30g/L

CONTACTS AND LOCATIONS:
Overall Officials: Wenhu Liu, doctor, Study Chair — Beijing Friendship Hospital; Zongli Diao, Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China